CLINICAL TRIAL: NCT01881295
Title: Bioavailability of Potassium From Potatoes and Potassium Gluconate
Acronym: Potato
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1301013174
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Potassium Bioavailability; Blood Pressure
Keywords: Potassium; Potato; French Fries; Bioavailability; Blood Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (9):
- Placebo control (Placebo Comparator): Subjects will consume tablets containing no potassium in addition to a basal diet containing 2336 mg potassium
  Interventions: Dietary Supplement: Placebo control
- Low dose potassium gluconate (Experimental): Subjects will consume 720 mg potassium in the form of potassium gluconate tablets daily in addition to a basal diet containing 2336 mg potassium
  Interventions: Dietary Supplement: Low dose potassium gluconate
- Medium dose potassium gluconate (Experimental): Subjects will consume 1440 mg potassium in the form of potassium gluconate tablets daily in addition to a basal diet containing 2336 mg potassium
  Interventions: Dietary Supplement: Medium dose potassium gluconate
- High dose potassium gluconate (Experimental): Subjects will consume 2160 mg potassium in the form of potassium gluconate tablets daily in addition to a basal diet containing 2336 mg potassium
  Interventions: Dietary Supplement: High dose potassium gluconate
- Low dose potato (Experimental): Subjects will consume 720 mg potassium in the form of potato daily in addition to a basal diet containing 2336 mg potassium
  Interventions: Dietary Supplement: Low dose potato
- Medium dose potato (Experimental): Subjects will consume 1440 mg potassium in the form of potato daily in addition to a basal diet containing 2336 mg potassium
  Interventions: Dietary Supplement: Medium dose potato
- High dose potato (Experimental): Subjects will consume 2160 mg potassium in the form of potato daily in addition to a basal diet containing 2336 mg potassium
  Interventions: Dietary Supplement: High dose potato
- High dose French fries (Experimental): Subjects will consume 2160 mg potassium in the form of french fries daily in addition to a basal diet containing 2336 mg potassium
  Interventions: Dietary Supplement: High dose French fries
- Basal diet control (Experimental): Subjects will consume a basal diet containing 2336 mg potassium daily
  Interventions: Dietary Supplement: Basal diet control

INTERVENTIONS:
Dietary Supplement: Placebo control
  Arms: Placebo control
Dietary Supplement: Low dose potassium gluconate
  Arms: Low dose potassium gluconate
Dietary Supplement: Medium dose potassium gluconate
  Arms: Medium dose potassium gluconate
Dietary Supplement: High dose potassium gluconate
  Arms: High dose potassium gluconate
Dietary Supplement: Low dose potato
  Arms: Low dose potato
Dietary Supplement: Medium dose potato
  Arms: Medium dose potato
Dietary Supplement: High dose potato
  Arms: High dose potato
Dietary Supplement: High dose French fries
  Arms: High dose French fries
Dietary Supplement: Basal diet control
  Arms: Basal diet control

SUMMARY:
This study is designed to compare the effect of sources of potassium on uptake and the effect of potassium on blood pressure.

DETAILED DESCRIPTION:
The study will compare uptake of potassium from three different doses and sources; supplements (720, 1440 and 2160 mg) potatoes (720, 1440 and 2160 mg) or French fries (2160 mg).

During 9 phases, participants will consume a controlled diet with the supplements, potato or french fries (every other week for 5 days). On the 4th day, blood and urine samples will be taken to monitor potassium uptake and excretion. Measures of blood pressure will be analyzed at defined time points throughout the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Able to adhere to the visit schedule, protocol requirements and available to complete the study
* Normotensive men and women
* Aged 20-60 years
* BMI of 15-35

Exclusion Criteria:

* Medication to treat hypertension or hypotension
* Medication known to affect electrolyte metabolism or contain high levels of potassium or sodium
* smoke cigarettes or use illegal drugs
* Hypertension or hypotension
* Diseases known to affect potassium metabolism
* Pregnant
* Allergic to nuts

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Bioavailability of Potassium | 5 days
  After 4 days of acclimation to the supplementation, absorption of potassium will be measured.

SECONDARY OUTCOMES:
Blood Pressure Response to Potassium | 6 days
  Differences in blood pressure will be measured between levels of potassium consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Weaver, Ph.D., Principal Investigator — Purdue University; Berdine R Martin, Ph.D., Study Director — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Macdonald-Clarke CJ, Martin BR, McCabe LD, McCabe GP, Lachcik PJ, Wastney M, Weaver CM. Bioavailability of potassium from potatoes and potassium gluconate: a randomized dose response trial. Am J Clin Nutr. 2016 Aug;104(2):346-53. doi: 10.3945/ajcn.115.127225. Epub 2016 Jul 13. PMID 27413123